CLINICAL TRIAL: NCT02321475
Title: Non-interventional Prospective Observational Study to Describe EGB 761® (Tanakan®) Effectiveness in the Treatment of Patients of Middle Age and Younger With Psycho-emotional Symptoms, Added to Cognitive Disorders.
Brief Title: EGb 761® (Tanakan®) Effectiveness in the Treatment of Patients of Middle Age and Younger With Psycho-emotional Symptoms, Added to Cognitive Disorders
Acronym: TAYPES
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-38-00240-138
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Cognitive Disorders
Keywords: Psycho-emotional symptoms
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Ginkgo biloba extract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Psycho-emotional symptoms, added to cognitive disorders: Patients of middle age and younger with psycho-emotional symptoms, added to cognitive disorders.
  Interventions: Drug: EGb761®

INTERVENTIONS:
Drug: EGb761®
  Other Names: Tanakan®

SUMMARY:
The purpose of this study is to determine the effectiveness of EGb 761® (Tanakan®) in Russian patients of middle age and younger, suffering from psycho-emotional symptoms added to cognitive disorders based on the improvement of FAM test (feeling-healthy, activity, mood test) score.

ELIGIBILITY:
Inclusion Criteria:

* Patients who signed the Informed Consent for participation in the observational study before collection of any information
* Patients who complain of psycho-emotional disturbance (of any intensity)
* Men and women aged 18-45 years, who prescribed to receive Tanakan® for cognitive disorders

Exclusion Criteria:

* Presence of any contraindications listed in the Tanakan® local SmPC (hypersensitivity to any of the components of Tanakan®, pregnancy, lactation, erosive gastritis in acute phase, gastric ulcer and duodenum ulcer in acute phase, acute cerebrovascular accident, acute myocardial infarction, congenital galactosemia, lactase deficiency, glucose-galactose malabsorption, haemolysis)
* Presence of dementia (according to Diagnostic and Statistical Manual of Mental Disorders [DSM IV])
* Disturbance of usual activities of daily living (e.g. self-care)
* Patients taking antipsychotic drugs, antidepressants, tranquillisers and nootropic agents
* Presence of any severe disease or condition which could affect cognitive function (e.g. Parkinson disease, epilepsy, brain inflammatory disease, major depression, recent post-stroke condition, recent brain-trauma etc.);
* Presence of anxiety or depression according to the Hospital Anxiety and Depression Scale (11 points and more).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Middle-age or younger patients with cognitive disorders and psycho-emotional symptoms (principal diagnosis).
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2014-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with increase of total medium FAM test score ≥1 after 3 months treatment | 3 months
  The FAM test is a questionnaire using three subscales (i.e. General health, Activity, and Mood). Scores for each subscale range from 3 to -3 (where -3 is bad and 3 is good). The total for each subscale and arithmetical mean is calculated.

SECONDARY OUTCOMES:
Change from baseline of total medium FAM test score. | 3 months
  The FAM test is a questionnaire using three subscales (i.e. General health, Activity, and Mood). Scores for each subscale range from 3 to -3 (where -3 is bad and 3 is good). The total for each subscale and arithmetical mean is calculated.
Change from baseline of short-time verbal memory | 3 months
  Investigator to assess short-time verbal memory using a set 10-words recall test.
Change from baseline of attention | 3 months
  Attention assessed using a digit-symbol coding test. The digit symbol score is the percentage of correct symbols completed in 90 seconds.
Percentage of patients who answered "Completely satisfied", "Rather satisfied", "Neither satisfied nor dissatisfied", "Rather dissatisfied" or "Completely dissatisfied", when assessing their satisfaction with Tanakan® | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (2):
- Russia (2):
  - Russian National Research Medical University, Moscow
  - First Moscow State Medical University, Moscow